CLINICAL TRIAL: NCT01433367
Title: A Prospective Observational Study Evaluating the Performance of the CerPass® Total Disc Replacement in Patients With Single-Level Cervical Disc Disease
Brief Title: A Clinical Trial Evaluating a Total Disc Replacement in Patients With Cervical Disc Disease
Acronym: CerPass
Status: Terminated | Type: Observational
Why Stopped: Marketing of CE marked device has been discontinued.
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA-CP-0904
Record Dates: First submitted 2011-06-10; First posted 2011-09-13 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cervical Disc Disease
Keywords: total disc replacement; cervical disc disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CerPass® Total Disc Replacement
  Interventions: Device: CerPass® Total Disc Replacement

INTERVENTIONS:
Device: CerPass® Total Disc Replacement — Single level cervical disc disease

SUMMARY:
This study will be a non-randomized trial consisting of patients with single level (C3 to C7) symptomatic cervical disc disease who have not previously received fusion surgery at the same level, and have failed to improve with conservative treatment for at least 6 weeks prior to enrollment, or who present with progressive neurological symptoms or signs in the face of conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

The criteria for inclusion into the proposed clinical study are as follows:

1. Age: 18-60 years of age (inclusive and skeletally mature);
2. A diagnosis of symptomatic cervical disc disease, defined as image-confirmed pathology: herniated disc, spondylosis, and/or loss of disc height. Spondylosis is defined as image-confirmed disc desiccation, loss of disc height, bridging osteophytes, and/or uncovertebral arthrosis. Loss of disc height is specified as a measurement of at least 25 degrees less than an adjacent nonsymptomatic level, but with a minimum of 1mm height remaining;
3. Functional neurological deficit (i.e., exhibits at least one sign associated with cervical level to be treated, including abnormal reflex, decreased motor strength, abnormal dermatome sensitivity, or pain in a dermatomal distribution);
4. Symptomatic level is C3-4, C4-5, C5-6 or C6-7 (one level);
5. Preoperative Neck Disability Index (NDI) greater than 30 points (considered moderate disability; Vernon 1991);
6. Unresponsive to conservative treatment for more than 6 weeks, and/or exhibits progressive symptoms and/or signs of nerve root and/or spinal cord compression in the face of conservative treatment;
7. Not pregnant, nor interested in becoming pregnant within the follow-up period of the study;
8. Willing and able to comply with the requirements defined in the protocol for the duration of the study;
9. Signed and dated Informed Consent.

Exclusion Criteria:

Patients with the following characteristics will not be eligible for entry into the proposed study:

1. Prior cervical fusion, prior laminectomy (prior cervical laminotomy that has not violated the facets need not be excluded), and/or prior cervical facetectomy at the operative level;
2. Requiring surgical treatment that would leave the patient with a postoperative deficiency of the posterior elements;
3. Signal changes in the cord on preoperative T2-weighted MRI and/or clinically significant myelopathy which would be described as gait disturbance, loss of manual dexterity, or bowel or bladder incontinence/retention.
4. Radiographic signs of significant instability at operative level (greater than 3mm translation, greater than 11 degree rotation different from adjacent level);
5. Bridging osteophytes or motion < 3 degrees;
6. Radiographic confirmation of significant facet joint disease or degeneration;
7. Chronic neck or arm pain of unknown etiology;
8. Cervical fracture, anatomic anomaly, or deformity (e.g. ankylosing spondylitis, scoliosis) at the levels to which the prosthesis will be attached;
9. Severe spondylolisthesis (greater than grade 1);
10. Endocrine disorders or connective tissue diseases;
11. Rheumatoid arthritis or other autoimmune disease;
12. Progressive neuromuscular disease, e.g., muscular dystrophy, multiple sclerosis;
13. Chronic steroid users;
14. Taking any medications or drugs in doses that are known to potentially interfere with the bone metabolism or soft tissue healing, which may include (but is not limited to) the following: inhaled glucocorticoids for asthma, corticosteroids, thyroid hormones, blood thinners (heparin, warfarin), gonadotropin-releasing hormone agonists for prostate cancer treatment, contraceptive medroxyprogesterone, lithium for bi-polar disorder treatment, anticonvulsants, aluminum-containing antacids, tetracycline;
15. Osteoporosis to a degree that spinal instrumentation would be contraindicated (DEXA T-score less than or equal to -2.5; DEXA necessary only if patient exhibits risk factors for low bone mass as quantified in DEXA screening questionnaire);
16. Diabetes mellitus requiring insulin management;
17. Presence of metastases or active spinal tumor malignancy;
18. Body Mass Index (BMI) > 40;
19. Active local or systemic infection, including AIDS, hepatitis;
20. Having been enrolled in another investigational device study within the last 90 days;
21. Having had another cervical device implanted that would interfere with the surgical approach, study or control device, or follow-up evaluations;
22. Demonstrates 3 or more signs of nonorganic behavior, such as Waddell's signs;
23. History of substance abuse;
24. Involved in spinal litigation;
25. Mentally incompetent;
26. Incarcerated.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Volunteers will be selected from the surgeon's existing clinic patients.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoints will be individual patient success at 24 months. | 24 months
  Success is defined as:
  Improvement in the Neck Disability Index (NDI) by ≥ 15 points at 24 months compared to Baseline;
  No device failures requiring revision, re-operation (including supplemental fixation), or removal from the patient;
  Maintenance or improvement of neurologic status (based on sensory, motor, and reflex assessment scores and observational gait analysis).

SECONDARY OUTCOMES:
Range of motion (ROM) | 24 months
  Range of Motion (ROM) defined as more than 3 degrees total flexion / extension. If the ROM is less than or equal to 3º the patient will be defined as having "non-motion."
SF-36 | 24-months
  SF-36 improvement of 15% at 24 months compared to Baseline
VAS analog pain scale (VAS) | 24-months
  Visual analog pain scale (VAS) improvement of 20 mm at 24 months compared to Baseline
Disc height improvement | 24-months
  Disc height from the lateral radiograph showing maintenance or improvement from baseline at 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Howell, Study Director — NuVasive
Locations (1):
- Hospital Del Prado, Tijuana, Estado de Baja California, Mexico